CLINICAL TRIAL: NCT01835899
Title: Safety, Tolerability and Pharmacokinetics of Multiple Rising Oral Doses of BI 1015550 Powder for Oral Solution in Healthy Male Volunteers q.d. or b.i.d.for 14 Days (a Randomised, Double-blind, Placebo-controlled Within Dose Groups Phase I Trial)
Brief Title: Safety, Tolerability and Pharmacokinetics of Multiple Rising Oral Doses of BI 1015550 Powder for Oral Solution
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1305.2; 2012-005614-19 (EudraCT Number: EudraCT)
Record Dates: First submitted 2013-04-09; First posted 2013-04-19 (Estimated); Results first posted 2016-01-22 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2015-12

CONDITIONS: Healthy
MeSH Terms: interventions — BI 1015550

ARMS (5):
- Placebo to BI 1015550 (Experimental): placebo
  Interventions: Drug: Placebo
- BI 1015550 low dose 1 (Experimental): powder for oral solution
  Interventions: Drug: BI 1015550
- BI 1015550 low dose 2 (Experimental): powder for oral solution
  Interventions: Drug: BI1015550
- BI 1015550 medium dose 1 (Experimental): powder for oral solution
  Interventions: Drug: BI 1015550
- BI 1015550 medium dose 2 (Experimental): powder for oral solution
  Interventions: Drug: BI 1015550

INTERVENTIONS:
Drug: Placebo — Placebo to BI 1015550
  Arms: Placebo to BI 1015550
Drug: BI 1015550 — medium dose 1 powder for oral solution
  Arms: BI 1015550 medium dose 1
Drug: BI 1015550 — medium dose 2 powder for oral solution
  Arms: BI 1015550 medium dose 2
Drug: BI1015550 — low dose 2 powder for oral solution
  Arms: BI 1015550 low dose 2
Drug: BI 1015550 — low dose 1 powder for oral solution
  Arms: BI 1015550 low dose 1

SUMMARY:
To investigate safety, tolerability, and pharmacokinetics of multiple rising oral doses of BI 1015550 in healthy male volunteers

ELIGIBILITY:
Inclusion criteria:

1. Healthy male subjects

Exclusion criteria:

1. Any relevant deviation from healthy conditions
2. Subjects unable to understand or to comply with study requirements

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1305.2.1 Boehringer Ingelheim Investigational Site, Mannheim, Germany

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study of multiple doses over 14 days was randomised, double-blind, and placebo-controlled within dose groups.
Groups:
- Placebo to BI 1015550: Subjects were orally administered twice daily with matching Placebo to BI 1015550 Powder for oral solution (PFOS), to have Volume identical to the active drug of the respective dose group.
- 1 mg BI 1015550: Subjects were orally administered twice daily with BI 1015550 1 mg PfOS (to have 4 mL volume of oral solution in total).
- 6 mg BI 1015550: Subjects were orally administered twice daily with BI 1015550 6 mg PfOS (to have 24 mL volume of oral solution in total).
Period: Overall Study
Arm/Group | Placebo to BI 1015550 | 1 mg BI 1015550 | 6 mg BI 1015550
Started | 6 | 9 | 9
Completed | 6 | 8 | 8
Not Completed | 0 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Other than stated above | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The treated set (TS) included all subjects who were dispensed study medication and were documented to have taken at least one dose of investigational treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo to BI 1015550 | 1 mg BI 1015550 | 6 mg BI 1015550 | Total
Number analyzed (Participants) | 6 | 9 | 9 | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.5 (9.9) | 38.7 (8.5) | 44.3 (8.3) | 42.0 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 6 | 9 | 9 | 24

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Drug-related Adverse Events
Description: Percentage of subjects with drug related Adverse events, as assessed by the investigator.
Time Frame: From first drug administration until last drug administration, upto 18 days.
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo to BI 1015550 | 1 mg BI 1015550 | 6 mg BI 1015550
Number analyzed (Participants) | 6 | 9 | 9
Percentage of participants | 16.7 | 44.4 | 11.1

2. Secondary Outcome: Cmax
Description: Maximum measured concentration of BI 1015550 in plasma.
Time Frame: 0:15h(hours); 0:30h; 0:45h; 1h;1:15h;1:30h; 2h;3h; 4h; 6h; 8h;10h; 12h; 24h; 34h and 47:55h after first drug administration.
Population: The PK analysis set (PKS) included all subjects of the TS who provided at least 1 observation for at least 1 secondary PK endpoint and who did not have a protocol violation relevant to the evaluation of PK.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | 1 mg BI 1015550 | 6 mg BI 1015550
Number analyzed (Participants) | 9 | 9
nmol/L | 24.0 (25.1) | 133.0 (14.9)

3. Secondary Outcome: AUCt,1
Description: Area under the concentration-time curve of BI 1015550 in plasma over a uniform dosing interval t after administration of the first dose
Time Frame: 0:15h(hours); 0:30h; 0:45h; 1h;1:15h;1:30h; 2h;3h; 4h; 6h; 8h;10h and 12h after first drug administration
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | 1 mg BI 1015550 | 6 mg BI 1015550
Number analyzed (Participants) | 9 | 9
nmol*h/L | 94.9 (10.3) | 622 (20.7)

4. Secondary Outcome: AUC0-infinity
Description: Area under the concentration-time curve of BI 1015550 in plasma over the time interval from 0 extrapolated to infinity.
Time Frame: as for outcome 2
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | 1 mg BI 1015550 | 6 mg BI 1015550
Number analyzed (Participants) | 9 | 9
nmol*h/L | 131 (18.6) | 958 (20.9)

5. Secondary Outcome: Cmax,ss
Description: Maximum measured concentration of BI 1015550 in plasma at steady state over a uniform dosing interval t.
Time Frame: 311:55h (hours); 312:15h; 312:30h; 312:45; 313h; 313:15h; 313:30h; 314h; 315h; 316h; 318h; 320h; 322h; 324h; 336h; 346h; 360h; 384h & 408h after first drug administration; last drug administration was at 312 h.
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | 1 mg BI 1015550 | 6 mg BI 1015550
Number analyzed (Participants) | 8 | 8
nmol/L | 28.6 (15.3) | 199 (14.5)

6. Secondary Outcome: AUCt,ss
Description: Area under the concentration-time curve of BI 1015550 in plasma at steady state over a uniform dosing interval t.
Time Frame: 311:55h; 312:15h; 312:30h; 312:45; 313h; 313:15h; 313:30h; 314h; 315h; 316h; 318h; 320h; 322h and 324h after first drug administration; last drug administration was at 312 h.
Population: PK set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | 1 mg BI 1015550 | 6 mg BI 1015550
Number analyzed (Participants) | 8 | 8
nmol*h/L | 148 (10.7) | 1090 (19.6)

ADVERSE EVENTS:
Time Frame: From first drug administration until last drug administration, upto 18 days.
Arm/Group | Placebo to BI 1015550 | 1 mg BI 1015550 | 6 mg BI 1015550
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 1/6 | 4/9 | 1/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo to BI 1015550 (N=6) | 1 mg BI 1015550 (N=9) | 6 mg BI 1015550 (N=9)
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
C-reactive protein increased (Investigations) | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 1 | 0

LIMITATIONS AND CAVEATS:
The study was prematurely completed as per protocol after 2 of the originally planned 4 dose groups ie., 1 mg BI 1015550 and 6 mg BI 1015550 because of higher than expected drug exposure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other